CLINICAL TRIAL: NCT04993924
Title: GnRH Antagonist Pre-treatment in the Early Follicular Phase for Resolution of a Baseline Functional Ovarian Cyst - A Proof-of-concept Pilot Study
Brief Title: GnRH Antagonist Pre-treatment in the Early Follicular Phase for Resolution of a Baseline Functional Ovarian Cyst
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Medical Center, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0024-21-ASF
Record Dates: First submitted 2021-02-20; First posted 2021-08-06 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: IVF; Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts | interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants (Experimental): Patients will start GnRH antagonist injections [Cetrotide (cetrolix) or Orgalutran (ganirelix) - depending on their primary prescription] for 3-6 days
  Interventions: Drug: Cetrorelix Acetate, Ganerelix Acetate

INTERVENTIONS:
Drug: Cetrorelix Acetate, Ganerelix Acetate — 3-6 days of 0.25 mg starting on day 2-3 of the menstrual cycle

SUMMARY:
In this study we would like to examine the effect of GnRH antagonist administration at the beginning of the follicular phase in patient presenting with a simple ovarian cyst 25-50 mm. The aim of this intervention is to allow a spontaneous regression of the ovarian cyst (if in nature) while ensuring a pituitary downregulation to prevent the beginning of a leading follicle recruitment. As previous studies using GnRH antagonist pre-treatment prior to GT initiation for other purposes demonstrated positive results (including different patient population) , no deleterious effects are expected.

DETAILED DESCRIPTION:
Reports on the effect of a baseline ovarian cyst on IVF cycle cancellation and outcome are scare and inconsistent. A cystic structure of the ovary may be functional or non-functional. Functional ovarian cysts are usually created by disruption of normal ovulation with the accumulation of intrafollicular fluid. Hormonal dysfunction prior to ovulation results in expansion of the follicular antrum with serous fluid. These cysts may be more frequent using Progesterone only contraceptives, Levonogetstrel-containing intrauterine device and following controlled ovarian stimulation during fertility treatments . Most functional cysts regress spontaneously within the first few days of menstruation or within the first 1-2 cycles and up to 6 months.

An ovarian cystic structure, even if hormonally inactive, may interfere with ovarian function during ovulation induction. These cysts may have a mechanical effect by reducing the space for growing follicles or by impairing ovarian blood supply. This may result in a lower number of oocytes and poor embryo quality, or utilization of higher doses of gonadotropins(GT) to reach the same oocyte yield.

Several studies have investigated the outcome of GnRH antagonist supplementation at the beginning of the menstrual cycle prior to GT stimulation mainly for the purpose of synchronization of antral follicles preventing a premature follicular recruitment. The delayed start protocol which combines estradiol priming followed by GnRH antagonist for 7 days at the beginning of menses prior to GT administration to further synchronize antral follicles improved ovarian response in poor responders and reduced cycle cancellation rate with no significant effect on pregnancy rates. A preliminary study investigated the effect of three day administration of GnRH antagonist at the beginning of the follicular phase prior to GT stimulation in normal responders regardless of baseline hormonal levels and found a trend towards increase in clinical pregnancy rate, and similar profiles of early embryo development, compared to standard fixed GnRH antagonist protocol.

Patients receiving an antagonist protocol usually start their stimulation on day 2-3 of menses. A baseline US and hormonal blood test are performed to determine adequacy of cycle start.

Patients presenting with a simple ovarian cyst larger then 25-30 mm in our unit, even in the presence of normal baseline estradiol levels are deferred to start their treatment in the following menstrual cycle as these structures may negatively affect treatment outcome. It is possible that these cystic structures, most being remnants of previous cycle, would have resolved spontaneously within a few days, but since GT treatment is to be started on the 2-3 day of the cycle to prevent leading follicle recruitment, we cannot wait to find out whether cyst has resolved and are inclined to postpone treatment to the following menstrual cycle.

Study aims: In this study we would like to examine the effect of GnRH antagonist administration at the beginning of the follicular phase in patient presenting with a simple ovarian cyst 25-50 mm. The aim of this intervention is to allow a spontaneous regression of the ovarian cyst (if in nature) while ensuring a pituitary downregulation to prevent the beginning of a leading follicle recruitment. As previous studies using GnRH antagonist pre-treatment prior to GT initiation for other purposes demonstrated positive results (including different patient population) , no deleterious effects are expected.

Materials and Methods: This is a proof-of-concept pilot study. Patients will be recruited at the reproductive medicine unit of Shamir Medical Center, Israel.

Study population: Patients undergoing controlled ovarian hyper stimulation at the IVF unit, Shamir medical center. Planned recruitment of 15 patients.

Sample size: This is a proof-of-concept pilot study to evaluate the feasibility and potential effectiveness of the intervention. A sample size of 15 patients will allow detecting the potential for use of cycles that would have been cancelled using standard protocols. As the comparator is mandatory cancellation, i.e. 0% use of cycles, this sample size is sufficient.

Study protocol:

Patients treated at the IVF unit at Shamir Medical Center planned for an antagonist cycle will undergo blood test and US exam at day 2-3 of their menstrual cycle. Patients will be recruited if a simple ovarian cyst > 25mm and < 50 mm is demonstrated upon US exam in the presence of E2 < 220 pmol/L. Following the initial US exam in the morning, if a simple cyst 25-50 mm will be demonstrated, the patient will receive a form explaining that her protocol may be changed according to blood test results with three possible options: 1. Continuation with the original protocol 2. Cancellation 3. Change in protocol as part of a research if she agrees to participate. As patients undergo blood draws in the morning, with results available in the afternoon, the initial recruitment will be performed over the phone with a verbal informed consent documented in the patients' medical file. A signed informed consent received at the following clinic visit.

Patients will receive a verbal explanation over the phone and following consent will start GnRH antagonist injections [Cetrotide (cetrolix) or Orgalutran (ganirelix) - depending on their primary prescription] for 3 days by which time a second blood test (for estradiol, progesterone, LH and FSH) and US exam will be performed.

* If cyst size has decreased to < 25 mm, and estradiol levels have remained < 220 pmol/L then GT stimulation will be started according to the original protocol.
* If cyst size has decreased in more than 10 mm mm but is still above 25mm, and estradiol levels have remained < 220 pmol/L additional 3 days treatment with Cetrotide (cetrolix) or Orgalutran (ganirelix) will be given.
* In case of no change/increase, the cycle will be cancelled. The patient will receive oral contraceptives for 2-3 weeks to time the next cycle and will start a new cycle once the current cyst resolves. The time to cyst resolution will be recorded.

When treatment is continued, the remnant of the cystic structure will be separately followed. Treatment outcomes will be recorded, including the number of follicles on both ovaries, number of mature oocytes of expected mature oocytes and number of embryos. Cystic outcome (if aspirated as part of the ovum pickup) will be recorded separately. In patients with a previous or a subsequent cycle with similar GT dosages, cycle outcomes will be compared to the cycle with the intervention.

Risks to subjects: No anticipated risks over regular stimulation protocol side effects.

Statistical analyses: Descriptive statistics will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Antagonist protocol.
2. Presentation for cycle initiation on day 2-3 of the menstrual cycle with a simple ovarian cyst >25 mm and < 50mm, and estradiol levels < 220 pmol/L.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Oocyte donor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Cyst resolution | 2 years
  Number of participants with a resolution/decrease in size of the cystic structure following GnRH antagonist.
Number of oocytes retrieved | 2 years
  cycle outcome - number of oocytes retrieved, of participants following the administration of the GnRH antagonist

SECONDARY OUTCOMES:
Number of patients which had an oocyte in the aspirated cystic content. | 2 years
  cystic content
Comparison of cycle outcome - oocyte number compared to a previous/future cycle cycle outcome compared to a previous cycle | 2 years
  Comparison to a similar cycle of the same patients using similar GT dosages - number of oocytes retrieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No